CLINICAL TRIAL: NCT02255812
Title: Taste Physiology in Healthy, Normal-weight Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: EKBB 289/12/2
Record Dates: First submitted 2014-08-06; First posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Exploratory Behavior
MeSH Terms: conditions — Exploratory Behavior | interventions — Citric Acid; Salts; Quinine; Sodium Glutamate; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 200 mL tap water (Placebo Comparator): Single intragastric instillation of 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 200 mL tap water via nasogastric tube
- 2 g citric acid (Active Comparator): Single intragastric instillation of 2 g citric acid in 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 2 g citric acid in 200 mL tap water via nasogastric tube
- 2 g salt (Active Comparator): Single intragastric instillation of 2 g salt in 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 2 g salt in 200 mL tap water via nasogastric tube
- 0.017 g quinine (Active Comparator): Single intragastric instillation of 0.017 g quinine in 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 0.017 g quinine in 200 mL tap water via nasogastric tube
- 1 g monosodium glutamate (Active Comparator): Single intragastric instillation of 1 g monosodium glutamate in 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 1 g monosodium glutamate in 200 mL tap water via nasogastric tube
- 25 g glucose (Active Comparator): Single intragastric instillation of 25 g glucose in 200 mL tap water via nasogastric tube
  Interventions: Dietary Supplement: Single intragastric instillation of 25 g glucose in 200 mL tap water via nasogastric tube

INTERVENTIONS:
Dietary Supplement: Single intragastric instillation of 200 mL tap water via nasogastric tube
  Arms: 200 mL tap water
Dietary Supplement: Single intragastric instillation of 2 g citric acid in 200 mL tap water via nasogastric tube
  Arms: 2 g citric acid
Dietary Supplement: Single intragastric instillation of 2 g salt in 200 mL tap water via nasogastric tube
  Arms: 2 g salt
Dietary Supplement: Single intragastric instillation of 0.017 g quinine in 200 mL tap water via nasogastric tube
  Arms: 0.017 g quinine
Dietary Supplement: Single intragastric instillation of 1 g monosodium glutamate in 200 mL tap water via nasogastric tube
  Arms: 1 g monosodium glutamate
Dietary Supplement: Single intragastric instillation of 25 g glucose in 200 mL tap water via nasogastric tube
  Arms: 25 g glucose

SUMMARY:
Taste physiology describes five main taste qualities in humans: sweet, sour, salty, umami and bitter. The receptors found on the tongue are also found in the entire gut. The correlation of stimulation of these gut receptors and brain activity has not yet been examined. The objectives are to investigate the effect of different taste substances on i) regional brain activity and ii) satiation peptide release.

ELIGIBILITY:
Inclusion Criteria:

* right-handed healthy males
* Body-mass index of < 25
* Age 18-45 years
* no drugs
* non-smoking

Exclusion Criteria:

* Smoking
* Substance abuse
* Regular intake of medications (except for oral contraceptives)
* Medical or psychiatric illness, especially: diabetes, pace-maker, claustrophobia
* History of gastrointestinal disorders
* Food allergies, glutamate intolerance
* Body piercings that cannot be removed

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
regional brain activity assessed by functional Magnetic Resonance Imaging (fMRI) | changes from baseline to one hour after treatment
  Changes in resting state functional connectivity

SECONDARY OUTCOMES:
gastrointestinal satiation peptide secretion | changes from baseline to one hour after treatment
  Unit of Measure: glucagon like peptide-1 (GLP-1) in pg/mL, peptide tyrosine tyrosine (PYY) in pg/mL and gastric inhibitory polypeptide (GIP) in pg/mL
glucose and insulin secretion | changes from baseline to one hour after treatment
  Unit of Measure: glucose in mmol/L, insulin in μU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland